CLINICAL TRIAL: NCT07062393
Title: Effect of Mobile Augmented Reality Counseling on Improving Shared Decision-Making in Thoracic Surgery: A Randomized Clinical Controlled Trial
Brief Title: Effect of Mobile Augmented Reality Counseling on Improving Shared Decision-Making in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chen Ying-Shian, MD, Tri-Service General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: TSGH-MAR-SDM-2025
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer Patients
Keywords: Shared decision making; Patient education; Augmented reality

STUDY DESIGN:
Intervention Model Description: This study employs a 2-period, 2-sequence crossover design in which all participants receive both interventions (traditional counseling and mobile augmented reality [MAR] counseling) in different sequences. Participants are randomly assigned to either the traditional-then-MAR group (T-M group) or the MAR-then-traditional group (M-T group). This design allows within-subject comparison of counseling effectiveness, minimizing individual variability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional First, Then MAR Counseling (T-M group) (Experimental): Participants receive traditional counseling first, followed by MAR counseling using a 3D mobile application.
  Interventions: Behavioral: Traditional Counseling → MAR Counseling
- MAR First, Then Traditional Counseling (M-T group) (Experimental): Participants receive MAR counseling first using a mobile 3D model app, followed by traditional counseling with CT images and verbal explanations.
  Interventions: Behavioral: MAR Counseling → Traditional Counseling

INTERVENTIONS:
Behavioral: Traditional Counseling → MAR Counseling — A single session begins with mobile augmented-reality counseling using interactive 3D models, followed by a standard verbal counseling with printed diagrams and CT images.
  Arms: Traditional First, Then MAR Counseling (T-M group)
Behavioral: MAR Counseling → Traditional Counseling — A single session begins with mobile augmented-reality counseling using interactive 3D models, followed by a standard verbal counseling with printed diagrams and CT images.
  Arms: MAR First, Then Traditional Counseling (M-T group)

SUMMARY:
This randomized clinical trial evaluates the effectiveness of Mobile Augmented Reality (MAR) counseling compared to traditional verbal counseling for patients undergoing thoracic surgery. MAR counseling integrates patient-specific 3D anatomical models to enhance understanding of surgical procedures and risks. The study assesses patient and caregiver satisfaction, decision-making confidence, and communication quality. Health care providers' perspectives on the counseling methods are also examined. Participants will be assigned to one of the two counseling groups and asked to complete a questionnaire immediately after the counseling session.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years and older
* Scheduled for elective thoracic surgery
* Able to understand written and spoken Mandarin
* Willing and able to provide informed consent
* Capable of completing questionnaires independently or with minimal assistance

Exclusion Criteria:

* Emergency surgery cases
* Severe cognitive impairment or psychiatric illness interfering with participation
* Visual or hearing impairments that prevent interaction with mobile devices
* Previous participation in a similar counseling trial
* Inability to complete follow-up procedures

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Shared decision-making score | Immediately after counseling session (single timepoint)
  Shared decision-making was evaluated using a validated questionnaire assessing patient perceptions of decision support, preparedness, and engagement. The total score ranges from 0 to 50, with higher scores indicating better shared decision-making.

SECONDARY OUTCOMES:
Patient counseling preference | Immediately after both counseling sessions
  Participants indicated their preference for either traditional counseling or MAR-based counseling after experiencing both, using a structured post-intervention questionnaire. The results were reported as percentages per group.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hsun Lin, MD, Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to ethical considerations and institutional policy. The informed consent obtained from participants does not include provisions for public data sharing.

REFERENCES:
- [Background] McDonald M, Shirk JD. The Effect of Digital Three-Dimensional Reality Models on Patient Counseling for Renal Masses. JSLS. 2023 Jan-Mar;27(1):e2022.00084. doi: 10.4293/JSLS.2022.00084. PMID 36818764
- [Background] Arjomandi Rad A, Vardanyan R, Thavarajasingam SG, Zubarevich A, Van den Eynde J, Sa MPBO, Zhigalov K, Sardiari Nia P, Ruhparwar A, Weymann A. Extended, virtual and augmented reality in thoracic surgery: a systematic review. Interact Cardiovasc Thorac Surg. 2022 Jan 18;34(2):201-211. doi: 10.1093/icvts/ivab241. PMID 34542639
- [Background] Deber RB, Kraetschmer N, Irvine J. What role do patients wish to play in treatment decision making? Arch Intern Med. 1996 Jul 8;156(13):1414-20. PMID 8678709
- [Background] Braddock CH 3rd, Fihn SD, Levinson W, Jonsen AR, Pearlman RA. How doctors and patients discuss routine clinical decisions. Informed decision making in the outpatient setting. J Gen Intern Med. 1997 Jun;12(6):339-45. doi: 10.1046/j.1525-1497.1997.00057.x. PMID 9192250
- [Background] Kessels RP. Patients' memory for medical information. J R Soc Med. 2003 May;96(5):219-22. doi: 10.1177/014107680309600504. No abstract available. PMID 12724430
- [Background] Lackey A, Donington JS. Surgical management of lung cancer. Semin Intervent Radiol. 2013 Jun;30(2):133-40. doi: 10.1055/s-0033-1342954. PMID 24436529
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Derived] Chen YS, Hsu YC, Romalee W, Wang DH, Lai J, Huang TW, Lin KH. Effect of Mobile Augmented Reality Counseling on Improving Shared Decision-Making in Thoracic Surgery: Randomized Clinical Crossover Trial. JMIR Mhealth Uhealth. 2025 Nov 13;13:e79632. doi: 10.2196/79632. PMID 41069141